CLINICAL TRIAL: NCT03832517
Title: A Phase 1, Double-Blind, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of RC-01 for Injection in Healthy Adult Subjects
Brief Title: Single and Multiple Dose Escalation Trial of an Intravenous Antibiotic RC-01
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: safety
Sponsor: Recida Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC-01-001
Record Dates: First submitted 2019-01-31; First posted 2019-02-06 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Single intravenous doses of RC-01 (Active Comparator): Single escalating doses of RC-01 from 200 mg to 1600 mg
  Interventions: Drug: Single intravenous doses of RC-01
- Single intravenous doses of placebo (Placebo Comparator): Single intravenous doses of placebo to match RC-01
  Interventions: Drug: Single intravenous doses of placebo
- Multiple intravenous doses of RC-01 (Active Comparator): Two or three times daily escalating intravenous doses of RC-01 for 10 days. Doses to be determined
  Interventions: Drug: Multiple intravenous doses of RC-01
- Multiple intravenous doses of placebo (Placebo Comparator): Two or three times daily intravenous doses of placebo to match RC-01
  Interventions: Drug: Multiple intravenous doses of placebo

INTERVENTIONS:
Drug: Single intravenous doses of RC-01 — Intravenous single escalating doses of RC-01
  Arms: Single intravenous doses of RC-01
Drug: Single intravenous doses of placebo — Intravenous single doses of placebo to match RC-01
  Arms: Single intravenous doses of placebo
Drug: Multiple intravenous doses of RC-01 — Multiple ascending doses of RC-01 given intravenously two or three times daily for 10 days
  Arms: Multiple intravenous doses of RC-01
Drug: Multiple intravenous doses of placebo — Multiple doses of placebo to match RC-01 given intravenously two or three times daily for 10 days
  Arms: Multiple intravenous doses of placebo

SUMMARY:
A Phase 1 study of the safety, tolerability and pharmacokinetics of a new antibiotic (RC-01). In Part 1 cohorts of healthy adults will participate in a single dose escalation study of increasing intravenous doses of RC-01. In Part 2 cohorts of healthy adults will participate in a multiple dose escalation study of increasing intravenous doses of RC-01 given either twice daily or three times daily.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Agrees to be available for all study visits and cooperate fully with the requirements of the study protocol, including the schedule of assessments
* Willing and able to provide written informed consent

Exclusion Criteria:

* Underlying hepatic, renal, metabolic, cardiovascular or immunologic disorders
* Unable to cooperate fully with the requirements of the study protocol, including the schedule of assessments, or likely to be non-compliant with any study requirements
* Women who are pregnant and/or nursing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-14 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with a treatment-related adverse event collected over the duration of the study | Up to the final follow-up 1 day visit
  Safety assessments will include physical examinations, vital signs including heart rate and respiratory rate, clinical laboratory tests (including hematology, serum chemistry, coagulation and urinalysis), and ECG parameters (including P-wave onset, QRS onset, QRS offset, and end of T wave)

SECONDARY OUTCOMES:
Plasma concentration time data for RC-01 and metabolites | Pre-dose through 24 hours after the final infusion of study drug
  Individual and mean plasma concentration time data for RC-01 and its metabolites
Bioavailability of RC-01 and other RC-01 metabolites | Pre-dose through 24 hours after the final infusion of study drug
  Levels of RC-01 and metabolites in blood
Elimination of RC-01 and its metabolites in the urine following single and multiple dose administration | Pre-dose through 24 hours after the final infusion of study drug
  Levels of RC-01 and its metabolites in the urine

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No